CLINICAL TRIAL: NCT01889381
Title: Human Craniomaxillofacial Allotransplantation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00067257
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Facial Injuries; Traumatic Wounds and Injuries; Craniofacial Injuries; Craniofacial Defects; Facial Transplantation; Facial Deformity
Keywords: Facial Injuries; Face Transplant; Facial Transplantation; Facial Deformity
MeSH Terms: conditions — Facial Injuries; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Transplantation) (Experimental): Face transplantation in combination with a novel donor bone marrow cell-based therapy followed by single-drug immunosuppression with potential weaning.
  Interventions: Drug: Bone marrow cell-based therapy & 1-drug immunosuppression.

INTERVENTIONS:
Drug: Bone marrow cell-based therapy & 1-drug immunosuppression. — This protocol uses a novel bone marrow cell-based therapy for composite tissue allotransplantation (CTA) rather than conventional triple-drug immunosuppression to facilitate long-term graft survival of deceased donor human faces under low-dose maintenance immunosuppression. Initial T-cell depletion with alemtuzumab is followed by upper extremity transplantation and tacrolimus maintenance therapy. Donor bone marrow cells are infused on Day 10 (±4 days) post-transplantation to elicit a host alloimmune response triggering exhaustion and deletion of the respective host (anti-donor) lymphocyte clones. Subsequently, tacrolimus therapy is given for at least 6 months before spaced weaning is considered in stable recipients.
  Other Names: Deceased donor face transplantation

SUMMARY:
Background: The human face is critically important for breathing, eating, seeing, and speaking/ communicating, but its most important job may be to look like a human face. Devastating facial deformities often cause affected individuals to avoid human contact and disappear from society. Although current surgical advancements can somewhat restore facial defects, this process often requires many operations and the resulting face only resembles the human face. To date, over 20 face transplants have been performed with highly encouraging functional and aesthetic results, but widespread clinical use has been limited due to the adverse effects of life-long and high-dose immunosuppression needed to prevent graft rejection. Risks include infection, cancer, and metabolic problems, all of which can greatly affect recipients' quality of life, make the procedure riskier, and jeopardize the potential benefits of face transplantation.

Study Design: This non-randomized, Phase II clinical trial will document the use of a new immunomodulatory protocol (aka - Pittsburgh Protocol, Starzl Protocol) for establishing face transplantation as a safe and effective reconstructive treatment for devastating injuries/ defects by minimizing maintenance immunosuppression therapy in face transplant patients. This protocol combines lymphocyte depletion with donor bone marrow cell infusion and has enabled graft survival using low doses of a single immunosuppressive drug followed by weaning of treatment. Initially designed for living-related solid organ donation, this regimen has been adapted for use with grafts donated by deceased donors. The investigators propose to perform 15 full or partial human face transplants employing this novel protocol.

Specific Aims: 1) To establish face transplantation as a safe and effective reconstructive strategy for the treatment of devastating facial injuries/defects; 2) To reduce the risk of rejection and enable allograft survival while minimizing the requirement for long-term, high-dose, multi-drug immunosuppression.

Significance of Research: Face transplantation could help injured individuals recover functionality, self-esteem, and the ability to reintegrate into family and social life as "whole" individuals. This protocol offers the potential for minimizing the morbidity of maintenance immunosuppression, thereby beneficially shifting the risk/benefit ratio of this life-enhancing procedure and enabling a wider clinical application of face transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Recent (≥6 months) or remote (i.e., several decades) craniomaxillofacial injury
* Male or female and of any race, color, or ethnicity.
* Aged 18-65 years.
* Strong desire to undergo craniomaxillofacial transplantation.
* Completes the protocol informed consent form.
* Non-smoker, defined by having never smoked or having quit >6 consecutive months prior to screening.
* No co-existing medical condition which, in the opinion of the study team, could affect the immunomodulatory protocol, surgical procedure, or functional results (see Exclusion Criteria below. If the condition is amenable to treatment, the study team must agree that said condition should not significantly enhance the surgical risks of full or partial craniomaxillofacial transplantation.)
* No co-existing psycho-social problems (i.e., alcoholism, drug abuse).
* Negative for malignancy for past 5 years.
* Negative for HIV at transplant.
* Negative crossmatch with donor.
* If female of child-bearing potential, negative serum pregnancy test.
* If female of child-bearing potential, consent to use reliable contraception for at least one year following transplantation.
* Consents to cell collection, storage, and bone marrow infusion as part of the treatment regime.
* USA citizen or equivalent.
* Patient agrees to comply with the protocol and states a dedication to the immunomodulatory treatment regime.

Exclusion Criteria:

* Positive for any of the following conditions:

  * Untreated sepsis.
  * HIV (active or seropositive).
  * Active tuberculosis.
  * Active Hepatitis B infection.
  * Hepatitis C.
  * Viral encephalitis.
  * Toxoplasmosis.
  * Malignancy (within past 5 years).
  * Current/recent (within 3 months of donation/screening consent) IV drug abuse.
  * Paralysis of ischemic, traumatic, or congenital origin.
  * Infectious, post infectious, or inflammatory (axonal or demyelinating) neuropathy.
  * Toxic neuropathy (i.e. heavy metal poisoning, drug toxicity, industrial agent exposure).
  * Mixed connective tissue disease.
* Conditions that, in the opinion of the study team, may impact the immunomodulatory protocol potentially exposing the recipient to an unacceptable risk under immunosuppressive treatment.
* A history of medical non-compliance.
* Sensitized recipients with high levels (50%) of panel-reactive Human Leukocyte Antigen (HLA) antibodies.
* Conditions that may impact the success of the surgical procedure or increase the risk of postoperative complications including inherited coagulopathies like Hemophilia, Von-Willebrand's disease, Protein C and S deficiency, Thrombocythemias, Thalassemias, Sickle Cell disease, etc.
* Mixed connective tissue diseases and collagen diseases can result in poor wound healing after surgery.
* Conditions that may impact functional outcomes including Lipopolysaccharidosis and amyloidosis (may impact nerve regeneration) or rare disorders of bone healing like osteopetrosis.
* Subjects with inadequate donor sites for autologous reconstruction in the event of post-transplant flap failure.
* Patients considered unsuitable per the consulted Psychiatric/ Psychologic appraisal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-08 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Graft Survival | Transplantation through end of study period (up to 5 years)
  Post-operative graft survival will be documented monthly Months 1-12 and quarterly (every 3 months) Years 2-5.

SECONDARY OUTCOMES:
Documentation of immunosuppression required by transplanted participants to maintain graft. | Transplantation to end of study period (up to 5 years)
  Post-operative serum trough levels will be documented daily Days 1-28, semiweekly Weeks 5-12, weekly Weeks 13-25, biweekly Weeks 26-38, monthly Months 10-12, and quarterly (every 3 months) Years 2-5.

CONTACTS AND LOCATIONS:
Overall Officials: Damon Cooney, MD, PHD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Background] Schneeberger S, Gorantla VS, Brandacher G, Zeevi A, Demetris AJ, Lunz JG, Metes DM, Donnenberg AD, Shores JT, Dimartini AF, Kiss JE, Imbriglia JE, Azari K, Goitz RJ, Manders EK, Nguyen VT, Cooney DS, Wachtman GS, Keith JD, Fletcher DR, Macedo C, Planinsic R, Losee JE, Shapiro R, Starzl TE, Lee WP. Upper-extremity transplantation using a cell-based protocol to minimize immunosuppression. Ann Surg. 2013 Feb;257(2):345-51. doi: 10.1097/SLA.0b013e31826d90bb. PMID 23001085